CLINICAL TRIAL: NCT02274155
Title: Phase Ib Study of a Monoclonal Antibody to OX40 (MEDI6469) Administered Prior to Definitive Surgical Resection Patients With Locoregionally Advanced, Oral Head and Neck Squamous Cell Carcinoma
Brief Title: Anti-OX40 Antibody in Head and Neck Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-042A
Record Dates: First submitted 2014-10-14; First posted 2014-10-24 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; anti-OX40 antibody; MEDI6469; Immunotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Anti-OX40 antibody administration 3 weeks prior to surgical resection
  Interventions: Drug: Anti-OX40 antibody administration; Procedure: Surgical Resection
- Group 2 (Experimental): Anti-OX40 antibody administration 2 weeks prior to surgical resection
  Interventions: Drug: Anti-OX40 antibody administration; Procedure: Surgical Resection
- Group 3 (Experimental): Anti-OX40 antibody administration 1 week prior to surgical resection
  Interventions: Drug: Anti-OX40 antibody administration; Procedure: Surgical Resection

INTERVENTIONS:
Drug: Anti-OX40 antibody administration — Anti-OX40 antibody administration at 0.4 mg/kg IV x 3 doses given on Days 1, 3 or 4, and 5 or 6 of study
  Other Names: MEDI6469
Procedure: Surgical Resection — Surgical Resection of Tumor

SUMMARY:
The purpose of this study is to test the safety of the anti-OX40 antibody, MEDI6469, given prior to surgery in patients with advanced head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
This phase Ib clinical trial uses MEDI6469 at various dose intervals prior to definitive surgical resection of patients with stage III and IV Oral Head and Neck Squamous Cell Carcinoma (OHNSCC) with the primary objective of determining the safety and feasibility of preoperative MEDI6469 administration. In addition, tumor tissue and peripheral blood will be obtained for exploratory immunologic end points including measurements of tumor infiltrating immune cell populations based on flow cytometry and immunohistochemistry as well as circulating immunological parameters that may correlate with changes induced by MEDI6469 administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with treatment naive, resectable, stage III or IV squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx who are candidates for definitive surgical resection followed by standard risk adapted adjuvant therapy.
* Histologic or cytologic diagnosis of a primary OHNSCC with no radiological evidence of metastatic disease is acceptable. Patients with bone or cartilage invasion and any T or N stage are acceptable.
* Patients with oral cavity primaries will be managed using conventional transoral or transcervical techniques; oropharynx or hypopharynx tumor will be managed with transoral robotic surgery; and larynx tumors (T3/T4 with thyroid cartilage invasion) will be managed by either total laryngectomy or larynx preservation surgery.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Laboratory values (performed within 28 days prior to enrollment) within protocol defined range
* Ability to give informed consent and comply with the protocol. Patients with a history of psychiatric illness must be judged able to understand the investigational nature of the study and the risks associated with the therapy.
* No active gastrointestinal bleeding.
* Anticipated lifespan greater than 12 weeks.

Exclusion Criteria:

* Locoregionally unresectable or Metastatic disease (stage IVB)
* Active infection.
* Active autoimmune disease including patients with Inflammatory Bowel Disease as determined by an autoimmune questionnaire.
* Previous treatment with mouse monoclonal antibodies
* Need for chronic maintenance oral steroids > 5mg prednisone daily equivalent.
* Any medical or psychiatric condition that in the opinion of the investigator would preclude compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2017-09-17 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility of definitive surgical resection for locoregionally advanced OHNSCC following MEDI6469 administration | 55 Days
  Patients will be seen in clinic 7 times over 55 days to identify any possible side effects or complications thought to be related to the study drug to help identify the optimal treatment schedule.

SECONDARY OUTCOMES:
Immunologic phenotypes of lymphocyte subsets | 55 days
  An uninvolved tumor-draining lymph node, primary tumor, and metastatic lymph nodes will be obtained during surgery, and peripheral blood will be collected 7 times over 55 days to identify the composition and immunologic phenotypes of lymphocyte subsets. This will also be compared to historical controls.

OTHER OUTCOMES:
Clinical Outcome of Imaging | 5 years
  Clinical surveillance for recurrence as per PET +/- CT within 6 months of completion of treatment exam. Clinical outcomes will be compared to historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B. Bell, MD, Principal Investigator — Providence Cancer Center
Locations (1):
- Portland Providence Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duhen R, Ballesteros-Merino C, Frye AK, Tran E, Rajamanickam V, Chang SC, Koguchi Y, Bifulco CB, Bernard B, Leidner RS, Curti BD, Fox BA, Urba WJ, Bell RB, Weinberg AD. Neoadjuvant anti-OX40 (MEDI6469) therapy in patients with head and neck squamous cell carcinoma activates and expands antigen-specific tumor-infiltrating T cells. Nat Commun. 2021 Feb 16;12(1):1047. doi: 10.1038/s41467-021-21383-1. PMID 33594075
- See also: Providence Cancer Center — http://oregon.providence.org/our-services/p/providence-cancer-center/